CLINICAL TRIAL: NCT02960594
Title: A Multi-center Study of hTERT Immunotherapy Alone or in Combination With IL-12 DNA Followed by Electroporation in Adults With Solid Tumors at High Risk of Relapse Post Definitive Surgery and Standard Therapy
Brief Title: hTERT Immunotherapy Alone or in Combination With IL-12 DNA Followed by Electroporation in Adults With Solid Tumors at High Risk of Relapse
Acronym: TRT-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Collaborators: University of Pennsylvania (Other); University of North Carolina (Other); Thomas Jefferson University (Other); University of Pittsburgh (Other); Barbara Ann Karmanos Cancer Institute (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TRT-001; NCT02327468 (obsolete NCT alias)
Record Dates: First submitted 2016-11-04; First posted 2016-11-09 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer; Lung Cancer; Pancreatic Cancer; Head and Neck Cancer; Ovarian Cancer; ColoRectal Cancer; Gastric Cancer; Esophageal Cancer; HepatoCellular Carcinoma
Keywords: Immunotherapy; Human Telomerase Reverse Transcriptase (hTERT); Breast Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; High Risk of Relapse; Post Definitive Surgery; Post Adjuvant Therapy; No Evidence of Disease
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Head and Neck Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Carcinoma, Hepatocellular | interventions — rocakinogene sifuplasmid; Interleukin-12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Arm 1 (Experimental): 2 mg INO-1400 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-1400
- Arm 2 (Experimental): 8 mg INO-1400 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-1400
- Arm 3 (Experimental): 2 mg INO-1400 + 0.5 mg INO-9012 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-1400; Biological: INO-9012
- Arm 4 (Experimental): 2 mg INO-1400 + 2 mg INO-9012 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-1400; Biological: INO-9012
- Arm 5 (Experimental): 8 mg INO-1400 + 0.5 mg INO-9012 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-1400; Biological: INO-9012
- Arm 6 (Experimental): 8 mg INO-1400 + 2 mg INO-9012 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-1400; Biological: INO-9012
- Arm 7 (Experimental): 2 mg INO-1401 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-1401
- Arm 8 (Experimental): 8 mg INO-1401 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-1401
- Arm 9 (Experimental): 8 mg INO-1401 + 0.5 mg INO-9012 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-9012; Biological: INO-1401
- Arm 10 (Experimental): 8 mg INO-1401 + 2 mg INO-9012 delivered intramuscularly followed by electroporation at Day 0, Weeks 4, 8, and 12
  Interventions: Biological: INO-9012; Biological: INO-1401

INTERVENTIONS:
Biological: INO-1400
  Other Names: hTERT
  Arms: Arm 1; Arm 2; Arm 3; Arm 4; Arm 5; Arm 6
Biological: INO-9012
  Other Names: IL-12
  Arms: Arm 10; Arm 3; Arm 4; Arm 5; Arm 6; Arm 9
Biological: INO-1401
  Other Names: SynCon TERT
  Arms: Arm 10; Arm 7; Arm 8; Arm 9

SUMMARY:
This is a Phase I, open label study to evaluate the safety, tolerability, and immunogenicity of INO-1400 or INO-1401 alone or in combination with INO-9012, delivered by electroporation in subjects with high-risk solid tumor cancer with no evidence of disease after surgery and standard therapy. Subjects will be enrolled into one of ten treatment arms. Subjects will be assessed according to standard of care. Restaging and imaging studies will be performed to assess disease relapse per NCCN guidelines. RECIST will be used to validate the findings in cases of relapse.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed and dated written IRB approved informed consent;
* 2. Males or females aged ≥18 years;
* 3. Subjects with breast, lung or pancreatic carcinoma who are at high risk of relapse post definitive therapy at least 4 and no more than 24 weeks from completion of definitive therapy at the time of signing informed consent as described below for each indication:

  * Breast carcinoma:
  * Lung carcinoma:
  * Pancreatic carcinoma:
  * Head and neck squamous cell carcinoma:
  * Ovarian cancer:
  * Colorectal cancer
  * Gastric and esophageal cancer
  * Hepatocellular carcinoma

Exclusion Criteria:

* 1. Previous treatment wth any TERT or IL-12 containing therapy, or any other DNA immunotherapy;
* 2. Any concurrent condition requiring the continued or anticipated use of systemic steroids (excluding non-systemic inhaled, topical skin and/or eye drop-containing corticosteroids) or immunosuppressive therapy (excludes low dose methotrexate). All other systemic corticosteroids must be discontinued at least 4 weeks prior to first Study Treatment;
* 3. Administration of any vaccine within 4 weeks of the first study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-12; Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Adverse events graded in accordance with "Common Terminology Criteria for Adverse Events (CTCAE)", NCI version 4.03 | Up to 2 years from first study treatment
Injection site reactions including, but not necessarily limited to, local skin erythema, induration, pain and tenderness at administration site | Up to 14 weeks
Changes in safety laboratory parameters | Up to 2 years from first study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vonderheide, MD, PhD, Principal Investigator — University of Pennsylvania; Autumn McRee, MD, Principal Investigator — University of North Carolina; Jennifer Johnson, MD, Principal Investigator — Thomas Jefferson University Hospitial; Anthony Shields, MD, Principal Investigator — Karmanos Cancer Center (Wayne State University); Nathan Bahary, MD, Principal Investigator — University of Pittsburgh; Ashish Chintakuntlawar, MBBS, PhD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (6):
- United States (6):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's Website — http://www.inovio.com